CLINICAL TRIAL: NCT00004661
Title: Study of the Regulation of Parathyroid Hormone Secretion in Pseudohypoparathyroidism
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11909; UCLA-541
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Pseudohypoparathyroidism
Keywords: endocrine disorders; pseudohypoparathyroidism; rare disease
MeSH Terms: conditions — Pseudohypoparathyroidism; Endocrine System Diseases; Rare Diseases

SUMMARY:
OBJECTIVES:

Determine the relationship between serum calcium concentrations and parathyroid hormone secretion in patients with pseudohypoparathyroidism.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients are tested for parathyroid hormone response following sequential graded intravenous infusions of sodium citrate and calcium gluconate. Assays include ionized calcium and intact parathyroid hormone.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Pseudohypoparathyroidism, i.e.: Renal resistance to parathyroid hormone OR Albright hereditary osteodystrophy No other illness unless related to pseudohypoparathyroidism No pregnant women

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1993-05

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell E. Geffner, Study Chair — University of California, Los Angeles